CLINICAL TRIAL: NCT01593371
Title: Comparing Effects of Metformin and Pioglitazone on Regulation of Serum Adipokines in Newly Diagnosed Type 2 Diabetes Patients
Brief Title: Comparison of Metformin and Pioglitazone Effects on Adipokines Concentrations in Newly Diagnosed Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Esteghamati, Professor Alireza Esteghamati, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 90-D-130-655
Record Dates: First submitted 2012-05-05; First posted 2012-05-08 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Adipokines; leptin; chemerin; omentin; metformin; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Active Comparator): patients receiving fixed dose metformin 1000 mg daily
  Interventions: Drug: Metformin
- Pioglitazone (Active Comparator): patients receiving fixed dose pioglitazone 30 mg daily
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Metformin — Metformin 1000 mg fixed dose, twice daily (500 mg tablets x 2)
  Arms: Metformin
Drug: Pioglitazone — Pioglitazone 30 mg fixed dose, twice daily (15 mg tablets x 2)
  Arms: Pioglitazone

SUMMARY:
Oral hypoglycemic agents encompass the mainstay of treatment in the majority of patients with type 2 diabetes. Thiazolidinediones (such a pioglitazone) and Biguanides (such as metformin), are two major groups of hypoglycemic medications that while function via different pathways, are both effective in short- and long-term glycemic control . These medications diminish or at least delay long term micro- and macrovascular complications associated with prolonged insulin resistance although at different rates. The mechanisms by which this aim is achieved, nevertheless, remains largely unclear. With adipokines playing a key role in development of both insulin resistance and atherosclerosis, oral hypoglycemic agents might regulate these substances by direct and indirect routes.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 2 diabetes patients based on American Diabetes Association criteria (2011) for diagnosis of diabetes

Exclusion Criteria:

* previous intake of oral hypoglycemic agents for treatment of diabetes or other hyperglycemia associated conditions
* intake of glucocorticoids in the past one year
* major illnesses of heart, lung, kidney, and liver.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of omentin | 12 weeks
  Serum concentrations of adipose tissue derived cytokine omentin
Serum concentrations of leptin | 12 weeks
  Serum concentrations of adipose tissue derived cytokine leptin

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Esteghamati, M.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Esteghamati A, Ghasemiesfe M, Mousavizadeh M, Noshad S, Nakhjavani M. Pioglitazone and metformin are equally effective in reduction of chemerin in patients with type 2 diabetes. J Diabetes Investig. 2014 May 4;5(3):327-32. doi: 10.1111/jdi.12157. Epub 2013 Oct 22. PMID 24843782